CLINICAL TRIAL: NCT02904031
Title: Randomized Phase II Study of First-Line FOLFOX Plus Panitumumab Versus 5FU Plus Panitumumab in RAS And BRAF Wild-Type Metastatic Colorectal Cancer Elderly Patients
Brief Title: Study of I Line FOLFOX + Panitumumab vs 5FU + Panitumumab in RAS and BRAF WT Metastatic Colorectal Cancer Elderly Patients
Acronym: PANDA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-003888-10
Record Dates: First submitted 2016-07-11; First posted 2016-09-16 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Elderly Metastatic Colorectal Cancer Patients
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Leucovorin; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFOX plus panitumumab (Experimental): * Panitumumab 6 mg/kg iv over 60 minutes, day 1; if the first infusion is tolerated, then subsequent infusions may be administered over 30 to 60 minutes;
  * Oxaliplatin 85 mg/sqm iv over 2 hours, day 1;
  * L-Leucovorin 200 mg/sqm iv over 2 hours, day 1;
  * 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. If no progression occurs, patients will receive maintenance panitumumab at the same dose used at the last cycle of the induction treatment. Panitumumab will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: 5-fluorouracil; Drug: oxaliplatin; Drug: l-leucovorin; Drug: panitumumab
- 5FU/LV plus panitumumab (Experimental): * Panitumumab 6 mg/kg iv over 60 minutes, day 1; if the first infusion is tolerated, then subsequent infusions may be administered over 30 to 60 minutes;
  * L-Leucovorin 200 mg/sqm iv over 2 hours, day 1;
  * 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. If no progression occurs, patients will receive maintenance panitumumab at the same dose used at the last cycle of the induction treatment. Panitumumab will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  Interventions: Drug: 5-fluorouracil; Drug: l-leucovorin; Drug: panitumumab

INTERVENTIONS:
Drug: 5-fluorouracil
Drug: oxaliplatin
  Arms: FOLFOX plus panitumumab
Drug: l-leucovorin
Drug: panitumumab

SUMMARY:
* Few data are available about the treatment of metastatic colorectal cancer (mCRC) elderly patients with anti-EGFR agents in combination with chemotherapy. Up today, most of the available data are from retrospective/post-hoc analyses, making them difficult to translate to everyday clinical practice.
* FOLFOX plus panitumumab is a standard first-line therapy option for RAS wild-type untreated mCRC patients. Slight adjustments in chemo-dosage are commonly applied in routinary practice to elderly patients, but those modified schedules have never been prospectively tested.
* In elderly patients, a reasonable upfront treatment is a fluoropyrimidine-based monotherapy plus bevacizumab, irrespectively of the molecular status of RAS.
* BRAF mutation is a strong negative prognostic factor associated to advanced age, poor performance status (PS), extended and aggressive disease and is associated to a lack of benefit from anti-EGFR moAb.
* Clinical definition of elderly (over 70 years old) CRC patients that may deserve a more or less intensive combination therapy is still debated. The cut-off of 75 years old combined with ECOG PS assessment is a reasonable approach for clearly defining candidates to different approaches31.
* Several geriatric screening tools have been used to identify patients with a geriatric profile potentially predicting for overall survival and risk of toxicity. The G8 screening tool has been validated in cancer patients showing the strongest prognostic value for overall survival; the CRASH score is able to stratify patients according an estimated risk of treatment-related toxicities.

On the basis of these considerations, the investigators designed the present randomized phase II trial of first-line therapy panitumumab in combination with simplified FOLFOX or with 5-fluorouracil, in previously untreated elderly patients with RAS and BRAF wild-type unresectable mCRC.

ELIGIBILITY:
Inclusion criteria

* Written informed consent to study procedures and to molecular analyses.
* Histologically proven diagnosis of colorectal cancer.
* Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
* At least one measurable lesion according to RECIST1.1 criteria.
* Availability of a tumoral sample (primary and/or metastatic sites).
* Age ≥ 70 years.
* ECOG PS 1 or 2 for patients aged 70 to 75 years; ECOG PS 0 or 1 for patients aged > 75 years.
* Life expectancy of at least 12 weeks.
* Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse.
* RAS and BRAF status wild-type of primary colorectal cancer or related metastasis, centrally assessed.
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥ 9 g/dl.
* Total bilirubin ≤ 1.5 time the upper-normal limits (UNL) of the normal values and ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases) alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases).
* Creatinine clearance ≥ 50 mL/min or serum creatinine ≤1.5 x UNL.
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception as approved by the investigator (barrier contraceptive measure or oral contraception).
* Geriatric assessment by means of G8 screening tool and CRASH score.
* Will and ability to comply with the protocol.

Exclusion criteria

* Previous treatment for metastatic disease.
* Radiotherapy to any site within 4 weeks before the study.
* Previous adjuvant oxaliplatin-containing chemotherapy.
* Previous treatment with EGFR inhibitors.
* Untreated brain metastases or spinal cord compression or primary brain tumors.
* History or evidence upon physical examination of CNS disease unless adequately treated.
* Symptomatic peripheral neuropathy > 1 grade NCIC-CTG criteria.
* Creatinine clearance < 50 mL/min or serum creatinine >1.5 x UNL.
* Clinical signs of malnutrition.
* Neutrophils <1.5 x 109/L, Platelets <100 x 109/L, Hgb <9 g/dl.
* Diagnosis of interstitial pneumonitis or pulmonary fibrosis.
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication.
* Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Definite contraindications for the use of corticosteroids and antihistamines as premedication.
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
* Sexually active males unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS). PFS is defined as the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first. | Up to 28 months
  July 2016 - November 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto IRCCS, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lonardi S, Rasola C, Lobefaro R, Rossini D, Formica V, Scartozzi M, Frassineti GL, Boscolo G, Cinieri S, Di Donato S, Pella N, Bergamo F, Raimondi A, Arnoldi E, Antonuzzo L, Granetto C, Zustovich F, Ronzoni M, Leo S, Morano F, Loupakis F, Buggin F, Zagonel V, Fassan M, Cremolini C, Boni L, Pietrantonio F; GONO Foundation Investigators. Initial Panitumumab Plus Fluorouracil, Leucovorin, and Oxaliplatin or Plus Fluorouracil and Leucovorin in Elderly Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer: The PANDA Trial by the GONO Foundation. J Clin Oncol. 2023 Dec 1;41(34):5263-5273. doi: 10.1200/JCO.23.00506. Epub 2023 Aug 3. PMID 37535876
- [Derived] Battaglin F, Schirripa M, Buggin F, Pietrantonio F, Morano F, Boscolo G, Tonini G, Lutrino ES, Lucchetti J, Salvatore L, Passardi A, Cremolini C, Arnoldi E, Scartozzi M, Pella N, Boni L, Bergamo F, Zagonel V, Loupakis F, Lonardi S. The PANDA study: a randomized phase II study of first-line FOLFOX plus panitumumab versus 5FU plus panitumumab in RAS and BRAF wild-type elderly metastatic colorectal cancer patients. BMC Cancer. 2018 Jan 25;18(1):98. doi: 10.1186/s12885-018-4001-x. PMID 29370781